CLINICAL TRIAL: NCT00473031
Title: Nutritional Regulation of Bone - Aim 1
Brief Title: The Effect of Weight Loss and Dietary Protein Intake on Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sue A. Shapses, Ph.D., RD, Professor, Rutgers University
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG0079; R01AG012161 (NIH); FP00011588 (Other Grant/Funding Number: Institute for the Advancement of Food and Nutrition Sciences)
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2022-01

CONDITIONS: Weight Loss; Bone Density
Keywords: bone mass; calcium absorption; bone quality; fracture risk
MeSH Terms: conditions — Weight Loss | interventions — Caloric Restriction; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): High Protein
  Interventions: Behavioral: Caloric restriction, high protein; Behavioral: Counseling
- 2 (Active Comparator): Normal Protein
  Interventions: Behavioral: Caloric restriction; normal protein; Behavioral: Counseling

INTERVENTIONS:
Behavioral: Caloric restriction, high protein — Weight loss with higher protein (35%) intake
  Arms: 1
Behavioral: Caloric restriction; normal protein — Weight loss with recommended level of protein (18%)intake
  Arms: 2
Behavioral: Counseling — Participants will be asked to attend eight 50-minute diet counseling sessions, with the opportunity to attend a total of approximately 28 diet counseling sessions, during the year.

SUMMARY:
The purpose of this study is to learn how the amount of protein during moderate weight loss influences bone health. We will also examine how two levels of protein intake affects diet quality.

DETAILED DESCRIPTION:
It is unclear whether protein intake during dieting influences bone density. This information is important for determining optimal nutrient requirements during weight loss. This study will compare the effects of weight loss with a lower-carbohydrate, high-protein (HP) diet to a high-carbohydrate, moderate protein (HC) diet on bone mass and quality in postmenopausal women (ages 50-70 years) with the hypothesis that bone turnover and loss of bone will be reduced on the HP compared to the HC weight loss diet. In a secondary aim, we will examine bone markers, hormones and the impact of protein intake on diet quality.

Participants will be randomly assigned to one of 2 groups: A) weight loss with recommended level of protein intake, and B) weight loss with higher protein intake. All participants will attend regular counseling sessions (about 50 minutes per session) with a dietitian for approximately 1 year, and will be asked to take a daily vitamin/mineral supplement. Also, depending on their usual food intake, they may be asked to take a calcium tablet to meet the recommended intake throughout the study period. Bone, mineral, protein and lipid markers, and hormones that influence bones will be measured. These measurements will provide information about body composition (fat, muscle mass, and bone mineral density). Participants will be asked to attend 8 diet counseling sessions, with the opportunity to attend a total of approximately 28 diet counseling sessions during the year.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women who are more than 2 years since last menses
* Obese or overweight
* Must live in the geographic vicinity of Rutgers University

Exclusion Criteria:

* Currently on any medication known to influence calcium or bone metabolism, including HRT, or with evidence of diseases known to influence calcium metabolism (i.e. metabolic bone disease, hyperparathyroidism, untreated thyroid disease, significant immune, hepatic, or renal disease, significant cardiac disease [i.e., heart attack or stroke in the past 6 months., abnormal EKG], active malignancy or cancer therapy within the past year)
* History of kidney stones
* Weight gain or weight loss (5% of body wt) within 3 months prior to recruitment
* Participation in other investigational studies during the 12-month study period
* Usually have a very high or low intake of calcium (more than 1500 or less than 500 mg per day)

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Changes in Bone density and quality | one year

SECONDARY OUTCOMES:
Changes in serum and urine bone markers, hormones, and proteins | one year
Nutrient Adequacy & Diet Quality with normal & higher protein intake | one year
  healthy eating index score

OTHER OUTCOMES:
Glomerular Filtration Rate with two levels of protein intake | one year
  GFR

CONTACTS AND LOCATIONS:
Overall Officials: Sue A. Shapses, PhD, Principal Investigator — Rutgers University, Nutritional Sciences
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

REFERENCES:
- [Background] Shapses SA, Riedt CS. Bone, body weight, and weight reduction: what are the concerns? J Nutr. 2006 Jun;136(6):1453-6. doi: 10.1093/jn/136.6.1453. PMID 16702302
- [Background] Riedt CS, Cifuentes M, Stahl T, Chowdhury HA, Schlussel Y, Shapses SA. Overweight postmenopausal women lose bone with moderate weight reduction and 1 g/day calcium intake. J Bone Miner Res. 2005 Mar;20(3):455-63. doi: 10.1359/JBMR.041132. Epub 2004 Nov 29. PMID 15746990
- [Background] Cifuentes M, Riedt CS, Brolin RE, Field MP, Sherrell RM, Shapses SA. Weight loss and calcium intake influence calcium absorption in overweight postmenopausal women. Am J Clin Nutr. 2004 Jul;80(1):123-30. doi: 10.1093/ajcn/80.1.123. PMID 15213038
- [Background] Goode LR, Brolin RE, Chowdhury HA, Shapses SA. Bone and gastric bypass surgery: effects of dietary calcium and vitamin D. Obes Res. 2004 Jan;12(1):40-7. doi: 10.1038/oby.2004.7. PMID 14742841
- [Result] Sukumar D, Ambia-Sobhan H, Zurfluh R, Schlussel Y, Stahl TJ, Gordon CL, Shapses SA. Areal and volumetric bone mineral density and geometry at two levels of protein intake during caloric restriction: a randomized, controlled trial. J Bone Miner Res. 2011 Jun;26(6):1339-48. doi: 10.1002/jbmr.318. PMID 21611972
- [Derived] Ogilvie AR, Schlussel Y, Sukumar D, Meng L, Shapses SA. Higher protein intake during caloric restriction improves diet quality and attenuates loss of lean body mass. Obesity (Silver Spring). 2022 Jul;30(7):1411-1419. doi: 10.1002/oby.23428. Epub 2022 May 11. PMID 35538903
- [Derived] Green CO, Badaloo AV, Hsu JW, Taylor-Bryan C, Reid M, Forrester T, Jahoor F. Effects of randomized supplementation of methionine or alanine on cysteine and glutathione production during the early phase of treatment of children with edematous malnutrition. Am J Clin Nutr. 2014 May;99(5):1052-8. doi: 10.3945/ajcn.113.062729. Epub 2014 Mar 5. PMID 24598154
- [Derived] Shapses SA, Sukumar D, Schneider SH, Schlussel Y, Sherrell RM, Field MP, Ambia-Sobhan H. Vitamin D supplementation and calcium absorption during caloric restriction: a randomized double-blind trial. Am J Clin Nutr. 2013 Mar;97(3):637-45. doi: 10.3945/ajcn.112.044909. Epub 2013 Jan 30. PMID 23364004